CLINICAL TRIAL: NCT07337642
Title: Comparing Collared and Collarless Femoral Stems in Total Hip Arthroplasty
Brief Title: Comparing Collared and Collarless Femoral Stems in Primary Total Hip Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00009612
Record Dates: First submitted 2026-01-09; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Primary Total Hip Arthroplasty

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Collard stem (Active Comparator)
  Interventions: Other: Collared Femoral Stem
- Collarless stem (Active Comparator)
  Interventions: Other: Collarless Femoral Stem

INTERVENTIONS:
Other: Collarless Femoral Stem — Patients will be randomized to one of two groups receiving either a collarless or collared femoral stem. Patients randomized to this group will receive a collarless femoral stem implant at time of surgery.
  Other Names: Collarless
  Arms: Collarless stem
Other: Collared Femoral Stem — Patients will be randomized to one of two groups receiving either a collarless or collared femoral stem. Patients randomized to this group will receive a collared femoral stem at the time of surgery.
  Other Names: collared
  Arms: Collard stem

SUMMARY:
This is a prospective randomized control trial comparing two collared and collarless femoral implants used in primary total hip arthroplasty. The specific aims of this trial are to:

SA1: Prospectively assess clinical outcomes in patients undergoing primary total hip arthroplasty with a collared versus collarless femoral stem of the same design.

SA2: Evaluate serial radiographs to quantify differences in subsidence between collared and collarless implant groups.

SA3: Report and compare incidence rates of intraoperative and postoperative periprosthetic fractures and aseptic loosening following primary total hip arthroplasty with use of either a collared or collarless stem.

Hypothesis: The addition of a collar to the same designed triple-taper primary hip stem will lead to a reduction in subsidence and incidence of perioperative and periprosthetic femur fractures.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years old) scheduled for primary, uncemented THA using a cementless femoral stem
* Diagnosis of primary osteoarthritis or other non-inflammatory degenerative joint disease.
* Ability and willingness to comply with study procedures and follow-up schedule.
* Ability to provide written informed consent

Exclusion Criteria:

* Patients not indicated for a cementless THA
* Prior surgery on the ipsilateral hip (e.g., prior THA, internal fixation, osteotomy)
* Use of cemented or hybrid femoral components.
* Revision THA or conversion THA
* Active or prior infection of the hip joint.
* Severe osteoporosis (T-score ≤ -2.5) or known metabolic bone disease.
* Inability to complete follow-up or anticipated relocation out of the area.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of femoral stem subsidence at 6 weeks, 6 months, and 1-year post-operation | 6 weeks, 6 months, and 1 year post operation
  Measurement of femoral stem subsidence at 6 weeks, 6 months, and 1-year post-operation used radiographic evidence.

CONTACTS AND LOCATIONS:
Locations (1):
- MedStar Georgetown University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-12-18): https://cdn.clinicaltrials.gov/large-docs/42/NCT07337642/Prot_000.pdf